CLINICAL TRIAL: NCT05206383
Title: Influence of Oral Messages on the Activity of Wrist and Finger Flexor Muscles - in the Context of Application of Sham Therapy
Brief Title: Influence of Oral Messages on the Activity of Wrist and Finger Flexor Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Paul II University in Biała Podlaska (Other)
Responsible Party: Principal Investigator, Kamil Zaworski, Director, John Paul II University in Biała Podlaska
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PopeJohnPaulIIStateSchHigherE3
Record Dates: First submitted 2021-12-28; First posted 2022-01-25 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Muscle; Communication; Activity, Motor
Keywords: muscle power; muscle activity; sham therapy; oral message
MeSH Terms: conditions — Communication; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study participants will be randomly qualified (allocated via a computer program) to the tree groups: A - positive message - placebo, B - negative message - nocebo, C - neutral message
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive message (Experimental): Group A - 30 subjects who will be told that positive message.
  Interventions: Behavioral: Positive message - placebo
- Negative message (Experimental): Group B - 30 subjects who will be told negative message.
  Interventions: Behavioral: Negative message - nocebo
- Neutral message (Experimental): Group C - 30 people who will be told neutral message.
  Interventions: Behavioral: Neutral message

INTERVENTIONS:
Behavioral: Positive message - placebo — Subjects who will be told that "the applied plastering method significantly increases muscle strength" (positive message - placebo).
  Arms: Positive message
Behavioral: Negative message - nocebo — Subjects who will be told that "the applied plastering method has no effect on muscle strength" (negative message - nocebo).
  Arms: Negative message
Behavioral: Neutral message — Subjects who will be told that "the applied plastering method is currently under investigation and the investigators do not know its effects" (neutral message).
  Arms: Neutral message

SUMMARY:
The aim of the study will be to evaluate the effect of oral messages on wrist and finger flexor muscle activity during the application of sham therapy in the form of paper plaster.

For years, research has been conducted on the effects of dynamic plaster and rigid plaster on muscle function. In many cases, reports from different authors are contradictory. Therefore, the planned study will use placebo paper plaster with no proven therapeutic effect.

DETAILED DESCRIPTION:
People's words can have a huge impact on how we interpret our surroundings, what we expect and experience, and how we behave. The placebo (and nocebo) effects are a clear example here. The way health professionals discuss, describe and inform patients about the characteristic effects of a given disease, its prevention, diagnosis and treatment influences patients' feelings and expectations, which in turn affects their psychobiological responses, subjective feelings and treatment outcomes.

The right choice of words by clinicians influences patients' response to medical treatments and procedures, both active and sham. The way in which information about the effects of treatment is communicated to patients can reinforce the outcomes of a particular treatment (placebo) or reverse clinically-proven effects of an active treatment, or even increase its adverse effects. The right messages can reduce the nocebo effect. And vice versa, the wrong choice of information provided may increase the patient's anxiety and disease symptoms.

The aim of the study will be to evaluate the effect of oral messages on wrist and finger flexor muscle activity during the application of sham therapy in the form of paper plaster.

Main hypothesis:

The use of a positive message will have an effect on increasing the activation and strength of the flexor muscles of the wrist joint and fingers.

Research questions:

1. Does a positive message have an effect on increasing the activation and strength of the flexor muscles of the wrist joint and fingers?
2. Does a negative message have an effect on increasing the activation and strength of the flexor muscles of the wrist joint and fingers? Does a neutral message have an effect on increasing the activation and strength of the flexor muscles of the wrist joint and fingers?

The study will be a prospective, flow-up study using a differential variable in the form of the type of message used (positive - placebo, negative - nocebo, neutral). The respondents will be randomly allocated to study groups using sealed allocation sheets.

Before taking part in the study, each subject will be familiarised with the course of the study and must give written informed consent to participate in the study and to be randomly assigned to a specific study group.

The subjects will be assessed twice - before applying a paper plaster and 10 minutes after applying the plaster and delivering a voice message.

ELIGIBILITY:
Inclusion Criteria:

* subjects not using non-steroidal anti-inflammatory drugs (NSAIDs) for at least one week prior to study entry,
* age - 19-24 years,
* written consent to participate in the study.

Exclusion Criteria:

* subjects studying for a degree in physiotherapy,
* subjects post surgery on the examined upper limb,
* subjects with past bone fractures in the examined upper limb,
* subjects who have had an injury to the examined upper limb within 6 months before the start of the study.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Dynamometer tests | Change in measured parameters 10 minutes after application of the plaster and delivery of the oral message relative to baseline measurement.
  Assessment of wrist and finger flexor muscle strength. Patient in sitting position with the elbow joint on the examined side bent and the forearm resting on the table. The patient squeezes the dynamometer for a period of 3-5 seconds.

SECONDARY OUTCOMES:
Testing with Naroxon Ultimum EMG | Change in measured parameters 10 minutes after application of the plaster and delivery of the oral message relative to baseline measurement.
  Assessment of wrist and finger flexor muscle activity. Patient in sitting position with the elbow joint on the examined side bent and the forearm resting on the table. The subject's arm is adducted, the wrist joint in an intermediate position. The electrodes are glued in the belly area of the flexor muscles of the wrist and fingers - about 2 cm from the medial epicondyle of the humerus in a distal direction at a distance of 1 cm from each other.
  The patient squeezes the dynamometer for a period of 3-5 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Zaworski, Study Chair — FIZJOPERFEKT Kamil Zaworski
Locations (1):
- Pope John Paul II State School Of Higher Education in Biała Podlaska, Biała Podlaska, Poland

IPD SHARING:
Plan to Share IPD: No